CLINICAL TRIAL: NCT05364034
Title: Effects of Urban Afforestation Activity on Thermal and Mechanical Pain Mechanisms: a Clinical Trial
Brief Title: Effects of Urban Afforestation Activity on Pain Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Mármol, Associate Professor, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AfforestPain
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: Green spaces; Nature-based activities; Horticultural therapy; Quantitative sensory testing; Pain mechanisms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urban Afforestation Group (Experimental): Participants will perform an afforestation activity with a duration of 90 minutes.
  Interventions: Other: Urban Afforestation Intervention Program

INTERVENTIONS:
Other: Urban Afforestation Intervention Program — An afforestation intervention program based on land cultivation and transplantation of several plants for 90 minutes will be implemented.
  Other Names: Nature-based activity; Afforestation activity

SUMMARY:
This single-group pretest-posttest clinical trial aims to evaluate the effects of a single-session afforestation activity on pain thresholds.

DETAILED DESCRIPTION:
Participants will perform an afforestation activity for a single session of 90 minutes. The therapist will direct the participants' attention to the visual, auditory, olfactory, and tactile features of the surrounding environment. A battery of quantitative sensory tests pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Free of pain in the hands, cheeks, lower back, wrists and trapezius muscles in the previous 3 months.
* Adults between 18 and 65 years.
* Any sex and gender.

Exclusion Criteria:

* Intake of any analgesic or psychotropic medication.
* Other severe or medically unstable diseases that may interfere with participation.
* Severe cognitive impairment (Mini-Mental State Examination score < 17 out of 30 points).
* Severe mental disorders in the acute phase or symptomatic phase.
* Severe intellectual disability.
* Behavioural alterations as this may interfere with their participation.
* Pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Cold pain detection threshold | Change from baseline cold pain detection threshold after 90 minutes.
  Cold pressor test will be employed (3±1°C). Participants will be instructed to submerge their nondominant hand in the cold water and report the initial occurrence of pain. Elapsed time in seconds will be recorded for the analysis as cold pain detection threshold. A cut-off time of 4 minutes is determined.
Cold pain tolerance threshold | Change from baseline cold pain tolerance threshold after 90 minutes.
  Cold pressor test will be employed (3±1°C). Participants will be instructed to submerge their nondominant hand in the cold water as long as they can endure the pain. Elapsed time in seconds will be recorded for the analysis as cold pain tolerance threshold. A cut-off time of 4 minutes is determined.
Cold pain intensity ratings | Change from baseline cold pain intensity ratings after 90 minutes.
  Cold pressor test will be employed (3±1°C). Cold pain intensities will be measured by asking the participants to report their maximal pain intensities by using the 101-point Numeric Rating Scale once the cold detection and tolerance thresholds are reached.
Wind-up ratio | Change from baseline wind-up ratio after 90 minutes.
  A response-dependent mechanical temporal summation method will be implemented by utilising a pinprick mechanical stimulator (256 mN). A single stimulus will be applied to the L2-L5 paraspinal muscles of the nondominant side and the participant will be asked to rate the pain intensity on the 101-point Numeric Rating Scale. After an interval of 10 seconds, a train of 10 stimuli will be applied on the same point with a mean cadence of 2 stimuli per second. This time the participant will be asked to rate the overall intensity of pain evoked by the stimuli series. The pain rating of the stimuli series will be divided by that of the single punctuation. This value will be recorded as the wind-up ratio.
Mechanical pain sensitivity | Change from baseline mechanical pain sensitivity after 90 minutes.
  The mechanical pain sensitivity of the participants' facial area will be assessed by using the same pinprick stimulator as for the wind-up ratio. A 2-sec pinprick stimulus will be applied on both cheeks three times. The interstimulus interval will be 10 seconds. Participants will be asked to rate the perceived pain intensity after each stimulus by using the 101-point Numeric Rating Scale. In case the participant does not report any pain, the minimum value of zero will be registered. A mean value of three measurements will be recorded as mechanical pain sensitivity.
Pressure pain detection thresholds | Change from baseline pressure pain detection threshold after 90 minutes.
  A hand-held dial pressure algometer device with the standard method of limits will be utilised. The application sites will consist of the muscle belly of the tibialis anterior and the middle of the dorsal aspect of the wrist joint line on the dominant side of participants. The patients will be asked to report the primary pain sensation to the evaluator. The value will be recorded in kg. A cut-off value of 1000 kPa is determined for safety reasons. A total of three measurements will be obtained at each site. Average of the second and third measurements will be recorded as pressure pain detection threshold.
Pressure pain intensity ratings | Change from baseline pressure pain intensity ratings after 90 minutes.
  The same instrument as in the pressure pain detection thresholds will be utilised. This time, nail of the dominant thumb will be subjected to two separate pressure levels, 294 kPa and 490 kPa, to obtain pressure pain intensity ratings. Upon reaching the aimed level, the pressure will be maintained for 2 seconds. Thereafter, participants will be asked to rate the evoked pain sensation by using the 101-point Numeric Rating Scale. Those who are unable to tolerate these pressure levels will be excluded from the analysis and handled as missing data. This procedure will be repeated three times. The average of the second and third measurements will be recorded as pressure pain ratings.
Pressure pain tolerance thresholds | Change from baseline pressure pain tolerance threshold after 90 minutes.
  The maximum pressure at which the participant defines the ongoing pain as intolerable is defined as the pressure pain tolerance threshold. A similar procedure as the detection thresholds will be adapted and followed this time for the mid-point of the upper border of the trapezius muscle and the nail cuticle of the ring finger on the nondominant side of participants. Average of the second and third measurements will be recorded as pressure pain tolerance threshold.

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel PÉREZ-MÁRMOL, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Granada, Faculty of Health Sciences, Granada, Spain

IPD SHARING:
Plan to Share IPD: No